CLINICAL TRIAL: NCT04123496
Title: Safety and Efficacy of an Accelerated Protocol of Intermittent Theta Burst Transcranial Magnetic Stimulation (TMS) to Enhance Performance and Promote Resilience in Astronauts: Study 1
Brief Title: rTMS to Enhance Cognitive Performance and Promote Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); The Translational Research Institute for Space Health (TRISH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00084982
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Cognition; Stress Reaction
Keywords: cognition; adult; prefrontal cortex; Transcranial Magnetic Stimulation; Stress, Psychological; memory; attention
MeSH Terms: conditions — Fractures, Stress; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (10):
- Dose 1 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is 5 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 2 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 2 is 10 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 3 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 3 is 15 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 4 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 4 is 20 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 5 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 5 is 25 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 6 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 6 is 30 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 7 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 7 is 35 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 8 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 8 is 40 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 9 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 9 is 45 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS
- Dose 10 (Experimental): All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 10 is 50 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Device: Repetitive Transcranial Magnetic Stimulation (rTMS) MagVenture MagPro TMS System would be utilized to deliver 3-minute sessions of intermittent theta burst to left dorsolateral prefrontal cortex.

SUMMARY:
The purpose of this study is to determine the most effective dose of brief, non-invasive brain stimulation (repetitive transcranial magnetic stimulation, rTMS) for improving cognitive functions such as attention and memory as well as to improve the ability to recover from stressful situations (stress resilience).

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) works by rapidly turning a focused magnetic field on-and-off repeatedly over your head, which passes directly through your hair, scalp, and skull and onto your brain, and can temporarily increase brain activity under the magnetic field. Repetitive transcranial magnetic stimulation (rTMS) is an FDA approved treatment for depression, and is used commonly to treat people for their depression. The rTMS treatment regime used in this study is different from the FDA approved treatment because you will receive up to ten treatments per day over five days instead of the FDA approved rTMS treatment regime of 25 treatments over 25 days. This sort of accelerated or high dose protocol has been shown to be safe and effective in the treatment of depression. We are hoping to find out if this treatment can be used as a treatment for improving cognitive function and stress resilience.

ELIGIBILITY:
Inclusion Criteria:

1. No history of mental or physical illness
2. No implanted metal in the body
3. College graduates (Associates degree or higher)
4. Negative urine pregnancy test, if female subject of childbearing potential
5. Able to read and understand questionnaires and informed consent

Exclusion Criteria:

1. Any current psychiatric diagnosis or current Clinical Global Impression ratings of psychiatric illness > 1
2. Current physical illness
3. History of CNS disease, concussion, overnight hospitalization, tumors, seizures, meningitis, encephalitis, abnormal CT/MRI of the brain
4. Moderate to severe traumatic brain injury (TBI)
5. History of a continuing significant laboratory finding
6. Frequent or severe headaches
7. Any history of psychotropic medication prior to study enrollment
8. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
9. active participation or plan for enrollment in another evidence-based clinical trial affecting psychosocial function
10. repeated abuse or dependence upon drugs (excluding nicotine and caffeine)
11. implanted devices/ferrous metal of any kind

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Roberts, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 2 | 3 | 2 | 0 | 2 | 2 | 21
  Male | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 1 | 2 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 3 | 4 | 3 | 4 | 2 | 3 | 3 | 2 | 4 | 31
  African American | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 5
  Other-Vietnamese American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other-Egyptian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Neurocognitive Performance (Fluid Cognition)
Description: Participants would complete a computerized batteries (Penn Computerized Neuropsychological Battery and NIH Cognition Battery). Tasks would assess the following domains: information-processing speed, executive function, sustained attention/vigilance, verbal memory, working-memory capacity, inhibition/impulsivity, and sensorimotor function. This composite includes all the tests noted above that are fluid ability measures: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. Higher values (positive changes from baseline) indicate better performance. The T-score has a mean of 50 in the general population and a SD of 10. Scores higher than the mean indicate better performance.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 63.500 (5.447) | 50.250 (10.079) | 59.750 (13.598) | 57.250 (13.150) | 60.500 (12.819) | 65.250 (5.795) | 58.250 (9.777) | 61.000 (3.464) | 70.333 (9.866) | 58.250 (4.856)

2. Primary Outcome: Change From Baseline in Neurocognitive Performance at 1 Week Post Treatment (Fluid Cognition)
Description: Participants would complete a computerized batteries (Penn Computerized Neuropsychological Battery and NIH Cognition Battery). Tasks would assess the following domains: information-processing speed, executive function, sustained attention/vigilance, verbal memory, working-memory capacity, inhibition/impulsivity, and sensorimotor function. This composite includes all the tests noted above that are fluid ability measures: Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. This composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. The T-score has a mean of 50 in the general population and a SD of 10. Scores higher than the mean indicate better performance.
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 72.500 (5.916) | 63.750 (5.852) | 67.750 (13.500) | 69.500 (11.790) | 70.000 (11.165) | 73.250 (5.252) | 71.000 (10.100) | 71.667 (5.508) | 69.000 (9.899) | 63.750 (7.588)

3. Primary Outcome: Change From Baseline in Neurocognitive Performance at 1 Month Post Treatment (Fluid Cognition)
Description: as for outcome 2
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 73.333 (9.292) | 65.000 (6.557) | 68.000 (11.106) | 71.250 (6.500) | 71.750 (7.762) | 68.333 (4.726) | 72.333 (10.263) | 74.000 (2.646) | 73.667 (3.215) | 67.500 (6.557)

4. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Connor Davidson Resilience Scale
Description: Participants would complete a series of questionnaires Connor Davidson Resilience Scale is a self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. The minimum value is a 0 and the maximum value is a 100. A higher score indicates higher resilience, which indicates a better outcome.
  -Questions are rated on a scale from 0-4, where a higher score reflects greater resilience.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dose 2; Dose 3; Dose 4; Dose 5; Dose 6; Dose 7; Dose 8; Dose 9; Dose 10: All participants will be randomized to one of 10 doses of accelerated rTMS. All doses are active and within established therapeutic levels of rTMS. Dose 1 is 5 sessions of 600 pulses at 120% of resting motor threshold. Intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds.
  rTMS: Device: Repetitive Transcranial Magnetic Stimulation (rTMS) MagVenture MagPro TMS System would be utilized to deliver 3-minute sessions of intermittent theta burst to left dorsolateral prefrontal cortex.
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 70.750 (10.079) | 74.250 (12.339) | 75.250 (12.842) | 80.000 (10.801) | 83.250 (7.274) | 72.750 (9.708) | 77.500 (5.447) | 85.333 (11.060) | 69.333 (19.630) | 74.250 (2.986)

5. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Perceived Stress Scale-10
Description: The investigators will use the Perceived Stress Scale 10 (PSS-10) to assess perceived stress using a 5-point Likert scale.
  Scoring Instructions: Total score is determined by adding together the scores of each of the four items. Questions 2 and 3 are reverse coded. Questions 1 and 4: 0 = Never; 1 = Almost never; 2 = Sometimes; 3 = Fairly often; 4 = Very often Questions 2 and 3: 4 = Never; 3 = Almost never; 2 = Sometimes; 1 = Fairly often; 0 = Very often.
  Scores range from 0 to 40 with higher scores indicating more stress.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 12.500 (3.109) | 12.500 (5.508) | 12.500 (4.796) | 9.750 (4.856) | 6.250 (5.909) | 11.500 (5.802) | 7.250 (5.560) | 8.667 (6.429) | 12.333 (6.658) | 11.250 (6.397)

6. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Inventory of Depression and Anxiety Symptoms-II
Description: The Inventory of Depression and Anxiety Symptoms-II (IDAS-II) is a 99-item self-report questionnaire assessing emotional and psychological symptoms across 18 subscales. Each item is rated on a 5-point Likert scale from 1 ("Not at all") to 5 ("Extremely").
  In this study, a composite score was calculated by summing responses across multiple relevant subscales (e.g., Dysphoria, Panic, Insomnia, Well-Being) to assess overall emotional distress and stress resilience.
  Minimum possible score: 99 (if all items scored 1) Maximum possible score: 495 (if all items scored 5) Higher scores indicate greater symptom severity and worse outcomes. Lower scores reflect better emotional functioning and greater resilience.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 136.250 (9.032) | 142.750 (18.209) | 144.500 (12.124) | 129.000 (10.520) | 127.750 (4.573) | 167.250 (47.594) | 133.500 (14.364) | 140.000 (22.650) | 136.667 (17.388) | 147.000 (25.534)

7. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Connor Davidson Resilience Scale
Description: The Connor Davidson Resilience Scale (CD-RISC 10) is a unidimensional self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. The minimum value is a 0 and the maximum value is a 100. A higher score indicates higher resilience, which indicates a better outcome.
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 72.000 (11.804) | 70.750 (7.848) | 76.000 (16.693) | 79.500 (9.678) | 80.000 (4.320) | 75.000 (7.024) | 84.000 (9.592) | 78.333 (15.044) | 69.000 (19.157) | 73.000 (7.958)

8. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Perceived Stress Scale-10
Description: as for outcome 5
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 15.500 (4.655) | 14.000 (2.449) | 10.000 (6.880) | 11.000 (4.082) | 6.750 (4.573) | 12.750 (3.594) | 6.750 (3.594) | 9.667 (7.234) | 13.667 (7.767) | 7.500 (2.646)

9. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Inventory of Depression and Anxiety Symptoms-II
Description: The Inventory of Depression and Anxiety Symptoms-II (IDAS-II) is a 99-item self-report questionnaire assessing emotional and psychological symptoms across 18 subscales. Each item is rated on a 5-point Likert scale from 1 ("Not at all") to 5 ("Extremely").
  In this study, a composite score was calculated by summing responses across multiple relevant subscales (e.g., Dysphoria, Panic, Insomnia, Well-Being) to assess overall emotional distress and stress resilience.
  Minimum possible score: 99 Maximum possible score: 495 Higher scores indicate greater symptom severity and worse outcomes. Lower scores reflect better emotional functioning and greater resilience.
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 142.750 (9.500) | 140.250 (12.500) | 140.750 (21.391) | 128.500 (14.617) | 125.250 (4.349) | 142.000 (22.672) | 135.750 (12.258) | 140.667 (24.786) | 133.333 (11.060) | 136.500 (18.083)

10. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Connor Davidson Resilience Scale
Description: as for outcome 7
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 69.000 (9.695) | 68.000 (17.795) | 80.000 (13.241) | 82.000 (12.702) | 84.500 (9.183) | 73.000 (7.303) | 81.500 (10.755) | 80.667 (16.042) | 68.667 (22.030) | 71.500 (5.196)

11. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Perceived Stress Scale-10
Description: as for outcome 5
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 13.000 (2.582) | 12.750 (2.986) | 8.250 (4.031) | 6.750 (4.787) | 5.250 (2.217) | 10.500 (6.856) | 9.250 (3.862) | 5.667 (7.371) | 13.000 (11.000) | 7.500 (2.646)

12. Secondary Outcome: Mean Score of Stress Resilience as Assessed by Inventory of Depression and Anxiety Symptoms-II
Description: as for outcome 9
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 140.250 (11.295) | 138.500 (17.311) | 142.750 (14.175) | 127.000 (10.551) | 122.500 (3.697) | 150.750 (31.879) | 134.250 (14.818) | 139.667 (21.127) | 128.667 (15.631) | 136.000 (15.100)

13. Secondary Outcome: Mean Score of Neurocognitive Performance (WINSCAT Composite)
Description: The WINSCAT battery includes 5 subtests: Code Substitution (CDS), Code Substitution Delayed Recognition (CDD), Delayed Matching to Sample (MSP), Mathematical Processing (MTH), and Running Memory Continuous Performance (CPT). Each subtest produces a standardized score (range: 0-100). Composite score is the sum of all subtests (range: 0-500). Higher scores indicate better cognitive performance. Baseline scores reflect initial neurocognitive status. WINSCAT assesses attention, memory, visual processing, and executive function.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 398.250 (70.415) | 302.500 (61.278) | 382.250 (41.428) | 366.250 (98.524) | 408.250 (71.481) | 367.750 (30.511) | 435.750 (14.569) | 382.000 (77.544) | 427.000 (17.088) | 400.750 (54.414)

14. Secondary Outcome: Mean Score of Neurocognitive Performance (WINSCAT Composite)
Description: The WINSCAT battery includes 5 subtests: Code Substitution (CDS), Code Substitution Delayed Recognition (CDD), Delayed Matching to Sample (MSP), Mathematical Processing (MTH), and Running Memory Continuous Performance (CPT). Each subtest produces a standardized score (range: 0-100). Composite score is the sum of all subtests (range: 0-500). Higher scores indicate better cognitive performance. This measure reflects post-treatment neurocognitive status following rTMS. Scores are compared to baseline to assess improvement. WINSCAT evaluates attention, memory, visual processing, and executive function.
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 406.750 (76.129) | 321.250 (28.028) | 388.250 (31.795) | 403.250 (74.813) | 445.000 (94.278) | 370.250 (18.554) | 459.000 (46.819) | 398.000 (11.358) | 503.667 (15.275) | 449.000 (46.275)

15. Secondary Outcome: Mean Score of Neurocognitive Performance (WINSCAT Composite)
Description: The WINSCAT battery includes 5 subtests: Code Substitution (CDS), Code Substitution Delayed Recognition (CDD), Delayed Matching to Sample (MSP), Mathematical Processing (MTH), and Running Memory Continuous Performance (CPT). Each subtest produces a standardized score (range: 0-100). Composite score is the sum of all subtests (range: 0-500). Higher scores indicate better cognitive performance. This measure reflects neurocognitive status 1 month after rTMS treatment. Scores are compared to baseline and 1-week post-treatment to assess sustained or enhanced cognitive improvement. WINSCAT evaluates attention, memory, visual processing, and executive function.
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 401.667 (75.646) | 380.333 (42.618) | 405.750 (50.328) | 414.750 (95.730) | 448.250 (55.883) | 424.500 (40.673) | 440.667 (26.312) | 431.667 (36.638) | 435.667 (62.405) | 429.250 (20.271)

16. Secondary Outcome: Mean Score of Neurocognitive Performance (Stress Total Score)
Description: is a 99-item self-report questionnaire assessing emotional and psychological symptoms across 18 subscales. For this outcome, a subset of items was used to assess stress resilience, likely drawn from the Well-Being or related subscales.
  Each item is rated on a 5-point Likert scale from 1 ("Not at all") to 5 ("Extremely"). Scores were summed across selected items.
  Minimum possible score: 0 Maximum possible score: 15 Lower scores indicate greater resilience and better emotional functioning. Higher scores indicate greater symptom severity and worse outcomes.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 12.500 (3.109) | 11.250 (6.702) | 13.500 (3.873) | 9.750 (4.856) | 6.250 (5.909) | 9.750 (6.602) | 9.750 (3.304) | 7.000 (7.937) | 13.333 (5.033) | 11.250 (6.397)

17. Secondary Outcome: Mean Score of Neurocognitive Performance (Stress Total Score)
Description: as for outcome 16
Time Frame: Post-treatment (within 1 week of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 15.500 (4.655) | 13.500 (3.109) | 11.500 (6.351) | 11.000 (4.082) | 6.750 (4.573) | 11.000 (5.354) | 11.500 (7.550) | 8.333 (8.505) | 14.000 (7.211) | 7.500 (2.646)

18. Secondary Outcome: Mean Score of Neurocognitive Performance (Stress Total Score)
Description: as for outcome 16
Time Frame: Post-treatment (within 1 month of completing rTMS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 4
score on a scale | 13.333 (3.055) | 11.000 (3.606) | 11.000 (3.367) | 6.750 (4.787) | 5.250 (2.217) | 7.750 (7.676) | 8.667 (6.028) | 7.000 (7.000) | 13.667 (10.017) | 7.500 (2.646)

ADVERSE EVENTS:
Time Frame: Participants were reviewed for adverse events from time of study entry (e.g., screening) to end of study (e.g., 1-month follow-up).
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Dose 10
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04123496/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04123496/ICF_000.pdf